CLINICAL TRIAL: NCT05804890
Title: Comparing Activated Carbon Cloth Dressing and Silver-Based Dressing in a Diabetic Foot Ulcer Population
Acronym: ZORFLEX
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National University of Malaysia (Other)
Collaborators: Dyamed Biotech Sdn Bhd (Unknown)
Responsible Party: Sponsor
Other Study IDs: FF-2022-294
Record Dates: First submitted 2022-12-07; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ZORFLEX: Activated Carbon Cloth Dressing
- AQUACEL: Silver-Based Dressing

SUMMARY:
One of the common complications of diabetes mellitus (DM) is Diabetic Foot Ulcer (DFU), which can subsequently lead to infections, gangrene, amputation or even death, if necessary care is not taken to curb with the condition. Despite the rapid advancements in the medical industry, diabetic foot ulcer (DFU) is considered as a major factor of morbidity and a leading cause of hospitalizations among diabetic patients. The risk of ulcer progression that may ultimately lead to amputation is elevated upon the development of DFU. It is estimated that DFU contributes approximately 50-70% of all lower limb amputations. In addition to rendering emotional and physical distress, DFU is also responsible for causing productivity and financial losses that lower the quality of life. The economic burden of the patients is further aggravated by the medical expenditure involved in the healing of DFU and/or lower extremity amputation. This study focuses on usage of a modern primary wound dressing in managing diabetic foot ulcer. The primary dressing used in this study is an activated carbon cloth dressing, which is applied directly to the wound bed and the "holes" in the net give access to the activated carbon which is made up of millions of micropores and within the walls of these micro pores, there is presence of electrostatic forces known as Van der Waals forces, which helps to trap and kill microorganisms such as MRSA and Pseudomonas aeruginosa. In addition, the dressings can regulate matrix metalloproteinases (MMPs) which are responsible for prolonged inflammation in chronic wounds like diabetic foot ulcers, and able to promote fibroblast migration and accelerate granulation tissue growth via its conductivity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Able and willing to provide consent and agree to comply with study procedures and follow-up evaluations
3. Patients with type 1 or type 2 diabetes mellitus.
4. Wagner classification grade 1-3
5. Patient's ulcer must be diabetic in origin. Debridement will be done prior to randomization.Ulcer size >1 and <25cm² ; ulcer duration of > 1 weeks
6. Additional wounds may be present but not within 3cm of the study wound.
7. Serum creatinine <3.0 mg/dl (266.0umol/L)
8. Glycosylated haemoglobin (HbA1c) <12%
9. Adequate circulation to the affected extremity as demonstrated by dorsum transcutaneousoxygen test (TcPO2) ≥ 30mmHg,ankle-brachial systolic index (ABSI) between 0.7 and 1.2 ortriphasic or biphasic Doppler arterial waveforms at the ankle of affected leg

Exclusion Criteria:

1. Unconfirmed Diabetes Mellitus diagnosis.
2. Wagner classification grade 4 and above.
3. Patients whose index diabetic foot ulcers are greater than 25cm² .
4. Patients considered not in reasonable metabolic control, confirmed by an HbA1c ≥ 12%within previous 90 days.
5. Patients whose serum creatinine levels are 3.0mg/dl or greater.
6. Patients with a known history of poor compliance with medical treatments.
7. Patients who have been previously randomized into this study, or are presentlyparticipating in another clinical trial.
8. Patients who are currently receiving radiation therapy or chemotherapy.
9. Patients with known or suspected local skin malignancy to the index diabetic ulcer.
10. Patients diagnosed with autoimmune connective tissues diseases.
11. Non-revascularizable surgical sites.
12. Any other pathology that would limit the blood supply and compromise healing
13. Patient who are pregnant or breast feeding.
14. Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Malaysian population diagnosed with diabetes mellitus type 2 with diabetic foot ulcer.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparing Activated Carbon Cloth Dressing and Silver-Based Dressing in a Diabetic Foot Ulcer Population. | 6 months
  The outcome measure is based on wound size in a span of 8 weeks. We used the same measurement tool for every patient's wound. The physiological parameters we use are FBC and CRP count. The questionnaires used was SF36.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Snyder RJ, Hanft JR. Diabetic foot ulcers--effects on QOL, costs, and mortality and the role of standard wound care and advanced-care therapies. Ostomy Wound Manage. 2009 Nov 1;55(11):28-38. PMID 19934461
- [Background] Shahbazian H, Yazdanpanah L, Latifi SM. Risk assessment of patients with diabetes for foot ulcers according to risk classification consensus of International Working Group on Diabetic Foot (IWGDF). Pak J Med Sci. 2013 May;29(3):730-4. doi: 10.12669/pjms.293.3473. PMID 24353617
- [Background] Aalaa M, Malazy OT, Sanjari M, Peimani M, Mohajeri-Tehrani M. Nurses' role in diabetic foot prevention and care; a review. J Diabetes Metab Disord. 2012 Nov 21;11(1):24. doi: 10.1186/2251-6581-11-24. PMID 23497582
- [Background] Iraj B, Khorvash F, Ebneshahidi A, Askari G. Prevention of diabetic foot ulcer. Int J Prev Med. 2013 Mar;4(3):373-6. No abstract available. PMID 23626896
- [Background] Fard AS, Esmaelzadeh M, Larijani B. Assessment and treatment of diabetic foot ulcer. Int J Clin Pract. 2007 Nov;61(11):1931-8. doi: 10.1111/j.1742-1241.2007.01534.x. PMID 17935551
- [Background] Leone S, Pascale R, Vitale M, Esposito S. [Epidemiology of diabetic foot]. Infez Med. 2012;20 Suppl 1:8-13. Italian. PMID 22982692
- [Background] Vileikyte L. Diabetic foot ulcers: a quality of life issue. Diabetes Metab Res Rev. 2001 Jul-Aug;17(4):246-9. doi: 10.1002/dmrr.216. PMID 11544609
- [Background] Murphy N. Reducing infection in chronic leg ulcers with an activated carbon cloth dressing. Br J Nurs. 2016 Jun 23;25(12):S38-44. doi: 10.12968/bjon.2016.25.12.S38. PMID 27345081
- [Background] Probst S, Saini C, Skinner MB. Comparison of sterile polyacrylate wound dressing with activated carbon cloth and a standard non-adhesive hydrocellular foam dressing with silver: a randomised controlled trial protocol. J Wound Care. 2019 Nov 2;28(11):722-728. doi: 10.12968/jowc.2019.28.11.722. PMID 31721666
- [Background] Scheer HS, Kaiser M, Zingg U. Results of directly applied activated carbon cloth in chronic wounds: a preliminary study. J Wound Care. 2017 Aug 2;26(8):476-481. doi: 10.12968/jowc.2017.26.8.476. PMID 28795884
- See also: Zorflex. 2017; https://tinyurl.com/yaoapvj8 (accessed 25 July 2017) — https://tinyurl.com/yaoapvj8